CLINICAL TRIAL: NCT01422096
Title: Effect of Short Term Ovarian Suppression on Androgen Overproduction in Overweight Girls With Androgen Excess (CBS007)
Brief Title: Effect of Short Term Ovarian Suppression on Androgen Overproduction in Overweight Girls With Androgen Excess
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study team decided not to pursue this study.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Assistant Professor of Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CBS007; CBS007 (Other: University of Virginia)
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Hyperandrogenemia; Obesity; Polycystic Ovary Syndrome
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- leuprolide (Experimental): leuprolide 11.25 mg IM with adrenal suppression/stimulation testing with dexamethasone/Cortrosyn and ovarian stimulation testing with r-hCG before and 3 weeks after injection
  Interventions: Drug: Leuprolide

INTERVENTIONS:
Drug: Leuprolide — depot leuprolide 11.25 mg if less than or equal to 37.5 kg or 15 mg if > 37.5 kg im once
  Other Names: Depot Lupron

SUMMARY:
This study will test whether short-term suppression of ovarian function can ameliorate androgen (male hormone) overproduction in overweight girls with androgen excess. The investigators hypothesize that one dose of depot leuprolide agonist administration will improve androgen levels in girls with ovarian androgen overproduction. Specifically, this intervention will improve androgen levels after ovarian stimulation testing with recombinant human chorionic gonadotropin (rhCG).

ELIGIBILITY:
Inclusion Criteria:

* overweight (>85th BMI%) females
* Early to late puberty (expected age range 7-18)
* Hyperandrogenemic (free testosterone greater than 2.5 standard deviations above the mean for normal control subjects of the same Tanner Stage)
* Screening labs within age-appropriate normal range, with the exception of a mildly low hematocrit (see below) and the hormonal abnormalities inherent in obesity which could include mildly elevated luteinizing hormone (LH), lipids, testosterone, prolactin, DHEAS, E2, glucose, and insulin and decreased follicle-stimulating hormone (FSH) and/or sex hormone-binding globulin (SHBG)

Exclusion Criteria:

* Screening labs outside of age-appropriate normal range
* Hemoglobin <12 mg/dL and hematocrit<36% (Subjects will be offered the opportunity to take iron supplementation for 60 days if their hematocrit is slightly low (33-36%) (suggestive of iron deficiency anemia) and will then return for retesting of their hemoglobin/hematocrit. If still <36%, they will be excluded.)
* Morning Cortisol <5 g/dL
* 17-hydroxyprogesterone >295 ng/dL
* History of Cushing's syndrome or adrenal insufficiency
* Pregnant

Ages: 7 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
17 hydroxyprogesterone responses to rhCG before and 4 weeks after depot leuprolide administration | 4 weeks after leuprolide

SECONDARY OUTCOMES:
Ovarian hormone precursor responses to rhCG before and 4 weeks after depot leuprolide administration | 4 weeks after leuprolide

CONTACTS AND LOCATIONS:
Overall Officials: Christine M. Burt Solorzano, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Research in Reproduction, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No